CLINICAL TRIAL: NCT02199600
Title: The Medacta International GMK Sphere Post-Marketing Surveillance Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02.014.01
Record Dates: First submitted 2014-07-07; First posted 2014-07-24 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Arthritis; Traumatic Arthritis; Rheumatoid Arthritis; Poly-arthritis; Avascular Necrosis
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GMK Sphere Knee Replacement (Other): Patients who comply with the protocol and received GMK Sphere component.
  Interventions: Device: GMK Sphere Knee Replacement

INTERVENTIONS:
Device: GMK Sphere Knee Replacement

SUMMARY:
This is a Post-Marketing Surveillance of GMK Sphere knee prosthesis.

DETAILED DESCRIPTION:
The clinical performance of the GMK® Sphere, manufactured by Medacta International, will be evaluated by a multicentre, prospective clinical surveillance study.

The Elective Orthopaedic Centre (EOC), in Epsom, Surrey, will be the study coordinating centre. Four further centres will participate in the clinical study, for five total centres. Each participating centre will recruit approximately 100 patients. Patient recruitment will cease when a cohort of 500 GMK® Sphere knee replacements have been implanted.

ELIGIBILITY:
Inclusion Criteria:

* A disabled or severely disabled joint as a result of arthritis, traumatic arthritis, rheumatoid arthritis, poly-arthritis or avascular necrosis
* Patients must be between the age of 18 and 80 at the time of consent
* Listed for total knee replacement surgery.
* Patients who are willing to give informed written consent

Exclusion Criteria:

* Progressive local or systemic infection
* Muscular loss, neuromuscular disease or vascular deficiency of the affected limb, making the operation unjustifiable
* Severe instability secondary to advance destruction of condylar structures or loss of integrity of the medial or lateral ligament
* Any patient who cannot or will not provide informed consent for participation in the study
* Those whose prospects for a recovery to independent mobility would be compromised by known coexistent, medical problems
* Patient whose BMI exceeds 40
* Any case not described in the inclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of the clinical outcome following total knee replacement using the Knee Society Score. | 6 months

SECONDARY OUTCOMES:
The OXFORD score as a measure of implant functionality. | pre-op, 6 months and annually for 10 years
Assessment of implant survivorship as a measure of safety and tolerability. | 6 weeks, 6 months, 3, 5, 7 and 10 years.
Radiographic analysis | pre-op, 6 months, 3, 5,7 and 10 years.
The EuroQol score as a measure of patient' quality of life. | pre-op, 6 months, 3, 5,7 and 10 years
Assessment of the clinical outcome following total knee replacement using the Knee Society Score | pre-op, at 6 months, at 3, 5, 7 and 10 years.

CONTACTS AND LOCATIONS:
Locations (4):
- AZ Maria Middelares, Ghent, Belgium
- United Kingdom (3):
  - Royal London Hospital, Whitechapel, London
  - Royal National Orthopaedic Hospital NHS Trust, Stanmore, Middlesex
  - The Elective Orthopaedic Centre (EOC), Epsom, Surrey